CLINICAL TRIAL: NCT03742960
Title: Sleep Subtypes in Adolescent Depression: Sleep Physiology and Treatment
Brief Title: Sleep Subtypes in Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University Hospital for Child and Adolescent Psychiatry and Psychotherapy Bern (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sleep Subtypes
Record Dates: First submitted 2018-10-31; First posted 2018-11-15 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Sleep Restriction (Experimental): Participants will be required to go to sleep half an hour later than their usual bedtime. Wake up time will be determined via their usual wake time.
  Interventions: Behavioral: Behavioral Sleep Restriction

INTERVENTIONS:
Behavioral: Behavioral Sleep Restriction — Participants will be instructed to go to bed 30 minutes later than their usual bedtime. On the other hand, wake up time will be unchanged resulting a nightly sleep restriction of 30 minutes. This protocol will be followed for two weeks.

SUMMARY:
The purpose of this study is to compare sleep neurophysiology and behavior in adolescents with MDD with hypersomnia (MDD-HYP) and insomnia (MDD-INS) with healthy controls (HC). In addition, the investigators will test the efficacy of a simple behavioral sleep restriction on mood and sleep in their sample.

DETAILED DESCRIPTION:
The World Health Organization has identified depression as the leading cause of burden of disease amongst young people. Subjective sleep complaints are often a core symptom of depression and highly prevalent with 60-90% of depressed adolescents suffering from disrupted sleep. This sleep disruption often takes the form of insomnia (e.g., difficulty falling or staying asleep, or waking too early) or hypersomnia (prolonged sleep episodes or excessive daytime sleepiness). The aim of the trial is to examine the efficacy of a simple behavioral sleep restriction two weeks in duration on mood and sleep in adolescents ages 14 to 17 years with and without major depressive disorder. During this period sleep is objectively measured using actigraphy and monitor mood using self-report. The results of the study will inform whether a simple behavioral sleep restriction beneficially impacts mood and sleep.

ELIGIBILITY:
Inclusion Criteria:

- This study will recruit adolescents (ages 14 to 17 years) with major depressive disorder (MDD) with insomnia (MDD-INS) and with hypersomnia (MDD-HYP) and age and gender matched controls (HC).

Inclusion Criteria:

Key inclusion criteria for MDD Hypersomnia Group:

* MDD as determined through the MINI-KID
* Determination of hypersomnia as defined by excessive daytime sleepiness, or long sleep duration.
* Written informed consent

Key inclusion criteria for MDD Insomnia Group:

* MDD as determined through the MINI-KID
* Determination of insomnia as defined by the insomnia severity index
* Written informed consent

Exclusion Criteria:

* Key exclusion criteria for all three groups include:

  * Current or lifetime experience of frank psychosis or mania
  * Presence of suicidal intent representing imminent risk as indicated during clinical interview
  * Medical or neurological condition that could impact brain functioning
  * History of physical brain injury or blow to the head resulting in loss of consciousness greater than 5 minutes
  * Do not meet criteria for substance or alcohol dependence in the last three months
  * Presence of an organic sleep disorder (e.g., narcolepsy, sleep apnea)

Additional exclusion criteria for healthy control group:

* Presence of psychiatric disorder
* Self-reported disrupted, short or ill-timed sleep

Additional exclusion criteria for MDD-INS and MDD-HYP:

• No sleep difficulties

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in self-reported sleep efficiency (defined as total sleep time divided by time in bed and thus expressed as a percentage) as assessed via sleep diary | Two weeks
  Changes in self-reported sleep efficiency will be measured via sleep diary. The data will be collected by ecological momentary assessment (EMA). Time in bed (TIB) is defined as the time between participants reporting going to bed and waking up. Total sleep time (TST) is defined as TIB minus the amount of time participants report taking to fall asleep (sleep onset latency; SOL) and the duration of waking after sleep onset (WASO).
Change in self-reported mood assessed via the Multidimensional Mood Questionnaire | Two weeks
  Changes in self-reported mood will be measured via ecological momentary assessment. Participants will fill out the Multidimensional Mood Questionnaire four times a day (morning, after school, at dusk and 30 minutes before bedtime). The Multidimensional Mood Questionnaire assesses the state "happy/sad" on a visual analog scale from 0 to 100. The mean across the day will be calculated.

SECONDARY OUTCOMES:
Change in Repetitive Negative Thinking (focus on problems) assessed by one question from the Response Style Questionnaire | Two weeks
  Change in repetitive negative thinking will be measured via ecological momentary assessment. Participants will answer the question about "focus on problems" on a scale from 0 [not at all] to 100 [very much]) once a day (evening).
Change in Repetitive Negative Thinking (focus on feelings) assessed by one question from the Response Style Questionnaire | Two weeks
  Participants will answer the question about "focus on feelings" on a scale from 0 [not at all] to 100 [very much]) once a day (evening).
Change in depressive symptoms from 1 to 3 days prior to the sleep manipulation and the end of the manipulation (second to last or last day of sleep manipulation) | Two weeks
  The change in depressive symptoms from 1 to 3 days prior to the sleep manipulation and the end of the manipulation (second to last or last day of sleep manipulation) will be measured via Center for Epidemiological Studies-Depression (CES-D; measures symptoms associated with depression), Strengths & Difficulties Questionnaires (SDQ; measures strengths and difficulties in general) and the Assessment of Snaith-Hamilton Pleasure Scale (SHAPS; assesses the presence of anhedonia [the inability to experience pleasure].
Change in anxiety symptoms from 1 to 3 days prior to the sleep manipulation and the end of the manipulation (second to last or last day of sleep manipulation) | Two weeks
  The change in depressive symptoms from 1 to 3 days prior to the sleep manipulation and the end of the manipulation (second to last or last day of sleep manipulation) will be measured via Screen for Child Anxiety-Related Emotional Disorders (SCARED; screens anxiety disorder categories).

CONTACTS AND LOCATIONS:
Overall Officials: Leila Tarokh, PhD, Principal Investigator — Universitätsklinik für Kinder- und Jugendpsychiatrie und Psychotherapie
Locations (1):
- Leila Tarokh, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided